CLINICAL TRIAL: NCT05480527
Title: Transcutaneous Pulsed Radiofrequency in Diabetic Neurophatic Pain
Brief Title: Transcutaneous Pulsed Radiofrequency in Diabetic Polyneuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, medical doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diabetic PNP
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-02

CONDITIONS: Neuropathy;Peripheral
Keywords: neuropathic pain; transcutaneous pulsed radiofrequency
MeSH Terms: conditions — Neuritis; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with bilateral neuropathic pain which treating active electrode (Active Comparator): 30 patients which treating with transcutaneous pulsed radiofrequency. All patients have diabetic polyneuropathy and confirmed with electroneuromyography.
  Interventions: Device: Transcutaneous pulsed radiofrequency current
- Patients with bilateral neuropathic pain which applied sham electrode (Sham Comparator): Sham electrodes will be applied to 30 patients. All patients have diabetic polyneuropathy and confirmed with electroneuromyography.
  Interventions: Device: Transcutaneous pulsed radiofrequency current

INTERVENTIONS:
Device: Transcutaneous pulsed radiofrequency current — Active treating group: 80 volts, 2Hz, 20 ms pulsed radiofrequency current will be applied to the tibial nerve trace in the ankle with electrodes. Sham group: Elelctrodes will be attached but radiofrequency current will not be applied.

SUMMARY:
Investigators want to investigate the efficacy of transcutaneous pulsed radiofrequency therapy in the treatment of diabetic peripheral neuropathy symptoms. For this purpose, investigators aimed to compare the results of two groups treated with sham electrode and active electrode.

DETAILED DESCRIPTION:
Peripheral neuropathic pain is common in diabetes mellitus. Distal symmetrical polyneuropathy is the most common form. These patients have complaints such as burning, freezing, tingling and pain in their hands and feet. Peripheral nerve blocks or sympathetic blocks are applied to patients who cannot be treated with medical agents.

Transcutaneous pulsed radiofrequency is a method used in the treatment of pain. The advantages of transcutaneous pulsed radiofrequency method are that it is not invasive, does not cause side effects, and does not interact with drugs. We want to investigate the efficacy of diabetic peripheral neuropathic pain treatment with this method.

Sixty diabetic polyneuropathy patients will be included in the study. Transcutaneous pulsed radiofrequency therapy with active electrode will be applied to half of the patients. Sham electrode will be used for the other half. Patients will not know which group they belong to. Two treatments will be applied with 7 days intervals. The duration of treatment will be 8 minutes.Each patient will receive a Leeds Assessment of Neuropathic Symptoms and Signs questionnaire (LANSS). Before the treatment, in the first month and third month after the treatment, the patients will be filled with a visual analog scale. The results between both groups will be statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes Mellitus
* Peripheric neuropathy with proved electroneuromyography

Exclusion Criteria:

* Additional endocrinological disease,
* Pregnancy, malignancy, motor deficit in lower extremities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baselina in pain on the Visual Analog Scale (VAS) at week 4 and 12 | Bseline, week 4 and week 12
  The visual analogue scale (VAS) is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain).

SECONDARY OUTCOMES:
Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | baseline, week4 and week 12
  it is a 7-item self-report scale developed to identify pain of predominantly neuropathic origin. Scores range 0 and 24. Scores of 12 and above are associated with neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Mehlika Panpallı Ateş, Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital; Damla Yürük, Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital; Ömer Taylan Akkaya, Study Director — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Dişkapi Reserch and Education Hospital, Ankara, Turkey (Türkiye)